CLINICAL TRIAL: NCT06660264
Title: Implementing Risk-Based Preemptive Pharmacogenomic (PGx) Testing in Employee Health
Brief Title: An Evaluation of the Impact of Pharmacist Personalized Medication Reviews With and Without a Discussion of Pharmacogenomic Results in an Employee Health Program.
Acronym: MyPGx
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Philip Empey, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY23050142
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Pharmacogenetics; Pharmacogenomic Drug Interaction
Keywords: Precision Medicine; Medication Review; PGx; Pharmacist; Pharmacogenomics; Employee health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Return of Pharmacogenomic Results (Other): Participants will be randomized to immediate versus delayed return of pharmacogenomic results obtained from testing conducted by an independent biobanking study (Pitt+Me Discovery). Participants in the immediate group will receive a pharmacist Personalized Medication Review with PGx results.
  Interventions: Other: Pharmacist Personalized Medication Review (PMR); Other: Discussion of Pharmacogenomic results during the PMR
- Delayed Return of Pharmacogenomic Results (Other): Participants will be randomized to immediate versus delayed return of pharmacogenomic results obtained from testing conducted by an independent biobanking study. Participants in the delayed group with receive a pharmacist Personalized Medication Review without PGx results. The delayed group will receive results from the independent biobanking study (Pitt+Me Discovery) at 12 months after the Personalized Medication Review.
  Interventions: Other: Pharmacist Personalized Medication Review (PMR)

INTERVENTIONS:
Other: Pharmacist Personalized Medication Review (PMR) — Pharmacist-provided review of current medications and assessment of potential medication related problems.
Other: Discussion of Pharmacogenomic results during the PMR — Return of pharmacogenomic results and discussion of impact on medications.
  Arms: Immediate Return of Pharmacogenomic Results

SUMMARY:
The goal of this prospective randomized clinical trial is to learn if a pharmacist-provided personalized medication review (PMR) that discusses pharmacogenomic test results will improve medication outcomes.

The primary aim is to identify patients within the Pitt/UPMC employee health programs who are most likely to benefit from PGx testing based on prescription history. The second aim is to determine the effect of the pharmacist-provided PMR including PGx test results.

Participants 18 years of age and older who have undergone PGx testing through a independent biobanking study (Pitt+Me Discovery) will be randomly assigned to receive PMR with a discussion of PGx test results or PMR without PGx results. Those who receive PMR only will receive PGx results one year after their PMR. Researchers will compare the groups to see if a pharmacist-provided PMR using PGx test results will lead to better medication outcomes and lower medical costs.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years old
* Enrolled in the UPMC insurance plan for at least 1 year
* Identified by UPMC Healthplan as a Pitt/UPMC employee who is likely to benefit from preemptive PGx panel testing based on polypharmacy, high annual prescription costs and a risk for poor medication-related outcomes based on exposure to medications with FDA or CPIC Level A/B PGx guidance using payer data
* Participating in Pitt+Me Discovery with elective return of PGx results

Exclusion Criteria:

* Previous panel PGx testing (self-reported)
* Have a terminal illness (specifically metastatic cancer, palliative care or hospice)
* Have had a liver, small bowel, or allogenic bone marrow/stem cell transplant
* Cannot provide informed consent and/or complete the study protocol due to serious cognitive impairment
* Institutionalized or too ill to participate (i.e. incarcerated, psychiatric or nursing home facility)
* Plan to drop UPMC Health Plan coverage for any reason within 12 months of enrollment
* Recent blood transfusion may be exclusionary only if the end of recruitment is nearing and there is insufficient time to observe a minimum waiting period between date of transfusion and date of sample collection. These minimum waiting periods are determined by type of transfusion: 7 days for platelets/plasma/cryoprecipitate; 2 months for packed red blood cells (PRBCs): and 6 months for whole blood or unknown type of transfusion. Although a transfusion is unlikely to have major effects on genotype results from a saliva sample, these time windows remove this concern.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Total Per Member Per Month (PMPM) Healthcare Costs | From 12 Months prior to PMR visit and from the PMR visit to 12 Months after the PMR visit
  Change in participant total per member/per month (PMPM) healthcare costs using healthplan claims data from 12 months prior to the pharmacist Personalized Medication Review (PMR) visit to 12 months after the PMR visit.

SECONDARY OUTCOMES:
Change in frequency of CPIC/FDA guideline concordant prescribing | Baseline, 12 Months after PMR visit
  Change in frequency of concordance of participant medication regimen with pharmacogenomics prescribing recommendations according to the Clinical Pharmacogenomics Implementation Consortium (CPIC) and U.S. Food & Drug Administration (FDA) guidelines using electronic health record data.
Change in healthcare utilization | From 12 Months prior to PMR visit and from the PMR visit to 12 Months after the PMR visit.
  Change in participant ER visits, hospitalizations, urgent care visits, specialist appointments, primary care appointments and unplanned care using UPMC Health Plan claims data from the year prior to the year after the pharmacist PMR visit.
Number of adverse events as assessed using the Patient-Reported Outcome Measure, Inquiry into Side-Effects (PROMISE) survey | 6 Months after PMR visit
  The Patient-Reported Outcome Measure, Inquiry into Side-Effects (PROMISE) allows participants to report common symptoms and suspected drug-related adverse events they may have experienced in the previous month. It includes a list of 22 common symptoms with option to write in other symptoms. For each symptom reported they are asked to indicate if they believe it might be a possible side effect of their medication. Scores range from 0 to 23. Higher scores indicate greater number of reported symptoms.
Change in Medication Access and Adherence Tool (MAAT) Score | Baseline, 6 Months after PMR
  The Medication Access and Adherence Tool (MAAT) will be used to assess change in medication adherence from Baseline to 6 Months. The MAAT is a tool that assesses participant-reported medication adherence. There are 5 questions with a score for each ranging from (1) not sure at all to (3) very sure. Possible scores range from 5 to 15, with higher scores indicating better medication adherence.
Health-systems Alliance for Integrated Medication Management (HAIMM) Score after Personalized Medication Review | After the PMR visit (up to 14 days after)
  The Health-systems Alliance for Integrated Medication Management (HAIMM) survey will be used to assess participant-reported understanding and satisfaction after the Personalized Medication Review session with the study pharmacist. The HAIMM contains 10 questions. Scores range from (0) not applicable to (4) strongly agree for 9 questions, and (1) poor to (5) excellent for the tenth question. Possible scores range from 4 to 41, with higher scores indicating greater participant satisfaction.
Health-systems Alliance for Integrated Medication Management (HAIMM) Score after Personalized Medication Review | 6 Months after PMR visit
  The Health-systems Alliance for Integrated Medication Management (HAIMM) survey will be used to assess participant-reported understanding and satisfaction after the Personalized Medication Review session with the study pharmacist. The HAIMM contains 10 questions. Scores range from (0) not applicable to (4) strongly agree for 9 questions, and (1) poor to (5) excellent for the tenth question. Possible scores range from 4 to 41, with higher scores indicating greater participant satisfaction.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, 6 Months after PMR visit
  The Patient-Reported Outcomes Measurement Information System (PROMIS) survey measures health across 7 domains including cognition, depression, fatigue, pain, physical fitness, sleep and social roles. The Promis Preference (PROPr) Utility Score will be used to combine 7 PROMIS domains into a single health utility score. There are 14 questions and responses range from (1) Not at all to (5) Very much. Scores range from 14 to 70, with higher scores indicating better general health.
Proportion of pharmacist recommendations were accepted | 12 months after PMR visit
  Proportion of pharmacist recommendations to address medication-related problems that were accepted by providers as assessed by EHR review.
Frequency of Actionable Genotypes | At 12 months after PMR visit
  Frequency of actionable genotypes (in the entire study population) based on report of a genotype-predicted phenotype. Actionable genotypes are defined as those with recommendations for a change in prescribing by a CPIC (Clinical Pharmacogenetics Implementation Consortium) guidelines or FDA recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Empey, PharmD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No